CLINICAL TRIAL: NCT03463447
Title: Measurement of Handgrip Strength and Pinch of Children and Adolescents Using an Electronic Dynamometer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Silvia Regina M. S. Boschi, PhD, University of Mogi das Cruzes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAAE: 67689517.7.0000.5497
Record Dates: First submitted 2018-03-06; First posted 2018-03-13 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Hand Strength
Keywords: Dynamometer; Handgrip; children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hand strength (Experimental): We selected volunteers without motor abnormalities with aged 6 to 17 years divided in groups (n = 30) according to an age group. The tests were performed in a single session lasting 20 minutes, when volunteers used a hydraulic dynamometer and an electronic dynamometer, in order to quantify the hand strength.
  Interventions: Device: Electronic Dynamometer; Device: Hydraulic dynamometer

INTERVENTIONS:
Device: Electronic Dynamometer — Mensuration of the handgrip strength of each volunteer using an electronic dynamometer.
Device: Hydraulic dynamometer — Mensuration of the handgrip strength of each volunteer using a hydraulic dynamometer.

SUMMARY:
This study has quantified the hand strength in movements of handgrip and pinch with electronic dynamometer.

DETAILED DESCRIPTION:
The hand is considered the most improved tool and differentiated of the human, with great importance in the accomplishment of numerous actions due to an essential function: The handgrip strength. The handgrip and pinch movements are very important for an accomplishment of daily activities. For an evaluation of the movements, the dynamometry has been used in many fields of health and frequently in the area of rehabilitation. However, if the type of dynamometer used is not suitable for children, a measurement of the handgrip may be compromised. Therefore, the present study verified the effectiveness of an electronic dynamometer to evaluate the handgrip strength and pinch in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* neurological disorder Absence
* Informed Consent signed by the responsible
* with preserved cognitive.
* consent form signed by the volunteer

Exclusion Criteria:

* change Absence of skeletal muscle in the upper limbs

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
Force | 15 minutes
  The force of handgrip, pinch pulp-side and pinch pulp-pulp movement. The test was measured 3 times with 1 minute interval . Unit of measurement: kilogram - force (kgf).

SECONDARY OUTCOMES:
Anthropometric variables (weight) | 1 minute
  weight of the volunteer. Unit of measurement: kilogram (Kg)
Anthropometric variables (height) | 1 minute
  height of the volunteer. Unit of measurement: meters (m)
Anthropometric variables (Measurements of the hands) | 3 minutes
  Measurements of the hands of each volunteer were evaluated. Unit of measurement: centimeters (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia R Boschi, PhD, Principal Investigator — University of Mogi das Cruzes
Locations (1):
- Silvia Regina Matos da Silva Boschi, Mogi das Cruzes, São Paulo, Brazil